CLINICAL TRIAL: NCT06286007
Title: Prevalence and Impact of Pertussis and RSV on Asthma Severity and Control
Acronym: PRIPASCO
Status: Recruiting | Type: Observational
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Collaborators: Translational Research In Airway Diseases Group (TRIAD) (Unknown); CIBER of Respiratory Diseases CIBERES (Unknown); Complexo Hospitalario Universitario de A Coruña (Other); Hospital de Galdakao (Other); Hospital Universitario Doctor Peset (Other); Hospital San Pedro de Alcantara (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Universitario Vall d´Hebron (Unknown); Universitat Autonoma de Barcelona (Other); Universidade de Santiago de Compostela (Unknown); Consortium for Biomedical Research in Epidemiology and Public Health (Unknown); Hospital Universitario Virgen del Rocio (Unknown); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); University Hospital Virgen de las Nieves (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Germans Trias i Pujol Hospital (Other); Hospital of Navarra (Other); Hospital Universitario de Jerez de la Frontera (Unknown); Hospital El Bierzo (Other); Hospital Clinico Universitario San Cecilio (Other); Hospital Donostia (Other); Hospital Universitario Central de Asturias (Other); Hospital Universitario de la Ribera (Unknown); Hospital Costa del Sol (Other); Hospital General Universitario Dr. Balmis (Unknown); Hospital de Sagunto (Other); Hospital Lluis Alcanyís de Xàtiva (Unknown); Hospital Universitario Lucus Augusti (Other); Hospital del Mar (Other); Hospital Universitario Virgen de la Arrixaca (Other); Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Francisco Javier González Barcala, Respiratory Medicine Specialist, Hospital Clinico Universitario de Santiago
Other Study IDs: PRIPASCO-2023
Record Dates: First submitted 2024-02-14; First posted 2024-02-29 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Asthma; Pertussis; RSV Infection
Keywords: Asthma; Pertussis; RSV Infection; Exacerbations
MeSH Terms: conditions — Asthma; Whooping Cough; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — The PCR samples (in all sites) and serology samples (yearly serology) in all the patients that are still included in the study will be obtained in each research centre and then sent to the coordinating centre
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PCR — Depending on the symptoms presented and date of symptom onset, for pertussis, patients will undergo a nasopharyngeal swab specimen for PCR if onset of the symptoms was within the past 3 weeks For RSV, patients will undergo a nasopharyngeal swab specimen for PCR if onset of the symptoms was within the past 72 hours.
  Other Names: Serology

SUMMARY:
The main objective is to estimate the annual symptomatic incidence of Bordetella pertussis and RSV infections in patients aged 18 years and over with asthma, which will be identified by PCR, for Bordetella pertussis and by PCR for RSV performed at a specific timepoint from onset of symptoms for each symptomatic Acute Respiratory Infection (ARI).

A multicentre prospective cohort study will be undertaken in Spain. Thirty-five centres from different autonomous communities in Spain will participate in the study.

Participants will be asked to report to the investigator if they experience an asthma exacerbation or symptoms of acute respiratory infection with 2 years follow up

DETAILED DESCRIPTION:
The main objective is to estimate the annual symptomatic incidence of Bordetella pertussis and RSV infections in patients aged 18 years and over with asthma, which will be identified by PCR, for Bordetella pertussis and by PCR for RSV performed at a specific timepoint from onset of symptoms for each symptomatic Acute Respiratory Infection (ARI).

A multicentre prospective cohort study will be undertaken in Spain. Thirty-five centres from different autonomous communities in Spain will participate in the study.

Participants will be asked to report to the investigator if they experience an asthma exacerbation or symptoms of acute respiratory infection with 2 years follow up

Depending on the symptoms presented and date of symptom onset, For pertussis, patients will undergo a nasopharyngeal swab specimen for PCR if onset of the symptoms was within the past 3 weeks For RSV, patients will undergo a nasopharyngeal swab specimen for PCR if onset of the symptoms was within the past 72 hours.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age 18 years and over)
* Diagnosed with asthma at least one year prior to the date of enrolment.
* Patients who, in the opinion of the investigator, can and will comply with the requirements of the study protocol for the duration of the follow-up period (e.g. agree to provide samples for testing, able to attend for testing upon asthma exacerbation and/or ARI symptoms occurring)
* Patients who are able to provide written informed consent.

Exclusion Criteria:

* Patients with a prior history of pertussis in the last 12 months
* Patients with ARI within the 2 weeks prior to enrolment
* Patients who have another respiratory disease other than asthma, alcohol or drug abuse at the time of being included in the study, or an active oncological disease (patients in treatment or follow-up for oncological disease) or pregnant women.
* Patients treated with immunosuppressive or immunomodulating agents not related to asthma diagnosis. will be excluded.
* Patients vaccinated for RSV will be also excluded (NOTE: -Patients that have received an RSV (investigational) vaccine or medicine for any of the above, should be excluded from the study from the beginning. Patients that might be vaccinated in the upcoming years, while the study is still ongoing, can enrol. However, from the moment they receive a vaccine, they should be excluded and no additional data will be collected. Data collected during the study up until the time of vaccination will still be included in the analysis).
* Patients vaccinated for B. Pertussis during the previous 12 months will be also excluded.
* Patients who plan to move during the study period will be excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adult patients (18 years and over) with asthma diagnosed at least one year before will be enrolled from the asthma clinics of selected hospitals.
  Every group (at each participating site) should include 35% of patients over 60 years old considering that this age-group has higher risk of infection and worse prognosis than the younger one.
Sampling Method: Non-Probability Sample
Enrollment: 784 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Bordetella pertussis and RSV infections in adult patients with asthma, | 2 years
  Incidence of Bordetella pertussis and RSV infections in adult patients with asthma,using PCR test

SECONDARY OUTCOMES:
To describe the seroprevalence of Bordetella pertussis in adult patients with asthma | 2 years
  To describe the seroprevalence of Bordetella pertussis in adult patients aged with asthma, at the time of inclusion, at 12 months, and at the end of two years follow-up, in all the patients that are still included in the study, using serological test
To describe the seroprevalence of RSV in adult patients with asthma | 2 years
  To describe the seroprevalence RSV in adult patients with asthma, at the time of inclusion, at 12 months, and at the end of two years follow-up, in all the patients that are still included in the study, using serological test
To evaluate the severity and control of the asthma caused by either BP or RSV infection | 2 years
  To evaluate, on an annual basis, the severity and control of the asthma, with regards to acute laboratory-confirmed respiratory illness caused by either BP or RSV infection during the study, using Asthma Control Test (ACT) questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Guiso N, Gallais JL, Gavazzi G, Pinquier D, Gaillat J. Incidence of pertussis in subjects aged 50years and older in France in 2013-2014. Med Mal Infect. 2018 Feb;48(1):30-36. doi: 10.1016/j.medmal.2017.09.002. Epub 2017 Oct 13. PMID 29037454
- [Background] Weinberger R, Riffelmann M, Kennerknecht N, Hulsse C, Littmann M, O'Brien J, von Kries R, von Konig CHW. Long-lasting cough in an adult German population: incidence, symptoms, and related pathogens. Eur J Clin Microbiol Infect Dis. 2018 Apr;37(4):665-672. doi: 10.1007/s10096-017-3158-6. Epub 2018 Jan 4. PMID 29302815
- [Background] Leong RNF, Wood JG, Liu B, McIntyre PB, Newall AT. High healthcare resource utilisation due to pertussis in Australian adults aged 65 years and over. Vaccine. 2020 Apr 23;38(19):3553-3559. doi: 10.1016/j.vaccine.2020.03.021. Epub 2020 Mar 24. PMID 32220516
- [Background] Mbayei SA, Faulkner A, Miner C, Edge K, Cruz V, Pena SA, Kudish K, Coleman J, Pradhan E, Thomas S, Martin S, Skoff TH. Severe Pertussis Infections in the United States, 2011-2015. Clin Infect Dis. 2019 Jul 2;69(2):218-226. doi: 10.1093/cid/ciy889. PMID 30321305
- [Background] Jenkins VA, Savic M, Kandeil W. Pertussis in high-risk groups: an overview of the past quarter-century. Hum Vaccin Immunother. 2020 Nov 1;16(11):2609-2617. doi: 10.1080/21645515.2020.1738168. Epub 2020 Apr 16. PMID 32298213
- [Background] Martinon-Torres F, Heininger U, Thomson A, Wirsing von Konig CH. Controlling pertussis: how can we do it? A focus on immunization. Expert Rev Vaccines. 2018 Apr;17(4):289-297. doi: 10.1080/14760584.2018.1445530. Epub 2018 Mar 12. PMID 29482390
- [Background] Martinón-Torres F. Expected and Unexpected Effects of Vaccination. In: Vesikari T, Van Damme P, editors. Pediatric Vaccines and Vaccinations, Cham (Switzerland): 2017, p. 3-13
- [Background] Aris E, Harrington L, Bhavsar A, Simeone JC, Ramond A, Papi A, Vogelmeier CF, Meszaros K, Lambrelli D, Mukherjee P. Burden of Pertussis in COPD: A Retrospective Database Study in England. COPD. 2021 Apr;18(2):157-169. doi: 10.1080/15412555.2021.1899155. Epub 2021 Apr 19. PMID 33866914
- [Background] Randi BA, Sejas ONE, Miyaji KT, Infante V, Lara AN, Ibrahim KY, Lopes MH, Sartori AMC. A systematic review of adult tetanus-diphtheria-acellular (Tdap) coverage among healthcare workers. Vaccine. 2019 Feb 14;37(8):1030-1037. doi: 10.1016/j.vaccine.2018.12.046. Epub 2019 Jan 7. PMID 30630694
- [Background] Rubin K, Glazer S. The pertussis hypothesis: Bordetella pertussis colonization in the etiology of asthma and diseases of allergic sensitization. Med Hypotheses. 2018 Nov;120:101-115. doi: 10.1016/j.mehy.2018.08.006. Epub 2018 Aug 10. PMID 30220328
- [Background] Martini H, Rodeghiero C, VAN DEN Poel C, Vincent M, Pierard D, Huygen K. Pertussis diagnosis in Belgium: results of the National Reference Centre for Bordetella anno 2015. Epidemiol Infect. 2017 Aug;145(11):2366-2373. doi: 10.1017/S0950268817001108. Epub 2017 Jun 5. PMID 28578723
- [Background] Marchi S, Montomoli E, Remarque EJ, Monteverde Spencer GT, Azzarello A, Viviani S, Trombetta CM. Pertussis over two decades: seroepidemiological study in a large population of the Siena Province, Tuscany Region, Central Italy. BMJ Open. 2019 Oct 30;9(10):e032987. doi: 10.1136/bmjopen-2019-032987. PMID 31666278
- [Background] Brugueras S, Rius C, Millet JP, Casals M, Cayla JA; Barcelona Pertussis Working Group. Does the economic recession influence the incidence of pertussis in a cosmopolitan European city? BMC Public Health. 2019 Feb 4;19(1):144. doi: 10.1186/s12889-019-6448-3. PMID 30717741
- [Background] Langsam D, Anis E, Haas EJ, Gosinov R, Yechezkel M, Grotto I, Shmueli E, Yamin D. Tdap vaccination during pregnancy interrupts a twenty-year increase in the incidence of pertussis. Vaccine. 2020 Mar 10;38(12):2700-2706. doi: 10.1016/j.vaccine.2020.01.095. Epub 2020 Feb 15. PMID 32070682
- [Background] Abu-Raya B, Maertens K, Edwards KM, Omer SB, Englund JA, Flanagan KL, Snape MD, Amirthalingam G, Leuridan E, Damme PV, Papaevangelou V, Launay O, Dagan R, Campins M, Cavaliere AF, Frusca T, Guidi S, O'Ryan M, Heininger U, Tan T, Alsuwaidi AR, Safadi MA, Vilca LM, Wanlapakorn N, Madhi SA, Giles ML, Prymula R, Ladhani S, Martinon-Torres F, Tan L, Michelin L, Scambia G, Principi N, Esposito S. Global Perspectives on Immunization During Pregnancy and Priorities for Future Research and Development: An International Consensus Statement. Front Immunol. 2020 Jun 24;11:1282. doi: 10.3389/fimmu.2020.01282. eCollection 2020. PMID 32670282
- [Background] Campins M, Moreno-Perez D, Gil-de Miguel A, Gonzalez-Romo F, Moraga-Llop FA, Aristegui-Fernandez J, Gonce-Mellgren A, Bayas JM, Salleras-Sanmarti L. [Whooping cough in Spain. Current epidemiology, prevention and control strategies. Recommendations by the Pertussis Working Group]. Enferm Infecc Microbiol Clin. 2013 Apr;31(4):240-53. doi: 10.1016/j.eimc.2012.12.011. Epub 2013 Feb 12. Spanish. PMID 23411362
- [Background] Redondo E, Rivero-Calle I, Mascaros E, Yuste JE, Fernandez-Prada M, Ocana D, Jimeno I, Gil A, Molina J, Diaz-Maroto JL, Linares M, Martinon-Torres F; en nombre de Neumoexpertos en Prevencion. [Vaccination against community acquired pneumonia in adults. Update 2021 of the position paper by Neumoexpertos en Prevencion Group]. Semergen. 2021 Sep;47(6):411-425. doi: 10.1016/j.semerg.2021.06.005. Epub 2021 Jul 29. Spanish. PMID 34332864
- [Background] Kandeil W, Atanasov P, Avramioti D, Fu J, Demarteau N, Li X. The burden of pertussis in older adults: what is the role of vaccination? A systematic literature review. Expert Rev Vaccines. 2019 May;18(5):439-455. doi: 10.1080/14760584.2019.1588727. Epub 2019 Mar 25. PMID 30887849
- [Background] Miyashita N, Akaike H, Teranishi H, Kawai Y, Ouchi K, Kato T, Hayashi T, Okimoto N. Diagnostic value of symptoms and laboratory data for pertussis in adolescent and adult patients. BMC Infect Dis. 2013 Mar 11;13:129. doi: 10.1186/1471-2334-13-129. PMID 23496900
- [Background] Schlaud M, Schmitz R, Poethko-Muller C, Kuhnert R. Vaccinations in the first year of life and risk of atopic disease - Results from the KiGGS study. Vaccine. 2017 Sep 12;35(38):5156-5162. doi: 10.1016/j.vaccine.2017.07.111. Epub 2017 Aug 8. PMID 28801155
- [Background] McDonald KL, Huq SI, Lix LM, Becker AB, Kozyrskyj AL. Delay in diphtheria, pertussis, tetanus vaccination is associated with a reduced risk of childhood asthma. J Allergy Clin Immunol. 2008 Mar;121(3):626-31. doi: 10.1016/j.jaci.2007.11.034. Epub 2008 Jan 18. PMID 18207561
- [Background] Vogt H, Braback L, Kling AM, Grunewald M, Nilsson L. Pertussis immunization in infancy and adolescent asthma medication. Pediatrics. 2014 Oct;134(4):721-8. doi: 10.1542/peds.2014-0723. Epub 2014 Sep 22. PMID 25246621
- [Background] Nagel G, Weinmayr G, Flohr C, Kleiner A, Strachan DP; ISAAC Phase Two Study Group. Association of pertussis and measles infections and immunizations with asthma and allergic sensitization in ISAAC Phase Two. Pediatr Allergy Immunol. 2012 Dec;23(8):737-46. doi: 10.1111/pai.12007. Epub 2012 Sep 24. PMID 23005697
- [Background] McKeever TM, Lewis SA, Smith C, Hubbard R. Vaccination and allergic disease: a birth cohort study. Am J Public Health. 2004 Jun;94(6):985-9. doi: 10.2105/ajph.94.6.985. PMID 15249303
- [Background] Buck PO, Meyers JL, Gordon LD, Parikh R, Kurosky SK, Davis KL. Economic burden of diagnosed pertussis among individuals with asthma or chronic obstructive pulmonary disease in the USA: an analysis of administrative claims. Epidemiol Infect. 2017 Jul;145(10):2109-2121. doi: 10.1017/S0950268817000887. Epub 2017 May 2. PMID 28462763
- [Background] Capili CR, Hettinger A, Rigelman-Hedberg N, Fink L, Boyce T, Lahr B, Juhn YJ. Increased risk of pertussis in patients with asthma. J Allergy Clin Immunol. 2012 Apr;129(4):957-63. doi: 10.1016/j.jaci.2011.11.020. Epub 2011 Dec 28. PMID 22206778
- [Background] Liu BC, McIntyre P, Kaldor JM, Quinn HE, Ridda I, Banks E. Pertussis in older adults: prospective study of risk factors and morbidity. Clin Infect Dis. 2012 Dec;55(11):1450-6. doi: 10.1093/cid/cis627. Epub 2012 Jul 17. PMID 22806592
- [Background] Harju TH, Leinonen M, Nokso-Koivisto J, Korhonen T, Raty R, He Q, Hovi T, Mertsola J, Bloigu A, Rytila P, Saikku P. Pathogenic bacteria and viruses in induced sputum or pharyngeal secretions of adults with stable asthma. Thorax. 2006 Jul;61(7):579-84. doi: 10.1136/thx.2005.056291. Epub 2006 Mar 3. PMID 16517571
- [Background] De Serres G, Shadmani R, Duval B, Boulianne N, Dery P, Douville Fradet M, Rochette L, Halperin SA. Morbidity of pertussis in adolescents and adults. J Infect Dis. 2000 Jul;182(1):174-9. doi: 10.1086/315648. Epub 2000 Jun 30. PMID 10882595
- [Background] Ristic M, Radosavljevic B, Stojanovic VD, Dilas M, Petrovic V. Performance of the new clinical case definitions of pertussis in pertussis suspected infection and other diagnoses similar to pertussis. PLoS One. 2018 Sep 20;13(9):e0204103. doi: 10.1371/journal.pone.0204103. eCollection 2018. PMID 30235311
- [Background] Wilkinson TMA, Van den Steen P, Cheuvart B, Baudson N, Dodet M, Turriani E, Harrington L, Meyer N, Rondini S, Taddei L, Mukherjee P. Seroprevalence of Bordetella pertussis Infection in Patients With Chronic Obstructive Pulmonary Disease in England: Analysis of the AERIS Cohort. COPD. 2021 Jun;18(3):341-348. doi: 10.1080/15412555.2021.1920904. Epub 2021 May 6. PMID 33955798
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Walsh EE. Respiratory Syncytial Virus Infection: An Illness for All Ages. Clin Chest Med. 2017 Mar;38(1):29-36. doi: 10.1016/j.ccm.2016.11.010. Epub 2016 Dec 27. PMID 28159159
- [Background] Matsumoto K, Inoue H. Viral infections in asthma and COPD. Respir Investig. 2014 Mar;52(2):92-100. doi: 10.1016/j.resinv.2013.08.005. Epub 2013 Sep 27. PMID 24636264
- [Background] Fleming DM, Taylor RJ, Lustig RL, Schuck-Paim C, Haguinet F, Webb DJ, Logie J, Matias G, Taylor S. Modelling estimates of the burden of Respiratory Syncytial virus infection in adults and the elderly in the United Kingdom. BMC Infect Dis. 2015 Oct 23;15:443. doi: 10.1186/s12879-015-1218-z. PMID 26497750
- [Background] Westerly BD, Peebles RS Jr. Respiratory syncytial virus infections in the adult asthmatic--mechanisms of host susceptibility and viral subversion. Immunol Allergy Clin North Am. 2010 Nov;30(4):523-39, vi-vii. doi: 10.1016/j.iac.2010.08.006. Epub 2010 Sep 22. PMID 21029936
- [Background] Falsey AR, Hennessey PA, Formica MA, Cox C, Walsh EE. Respiratory syncytial virus infection in elderly and high-risk adults. N Engl J Med. 2005 Apr 28;352(17):1749-59. doi: 10.1056/NEJMoa043951. PMID 15858184
- [Background] Falsey AR, Walsh EE, Capellan J, Gravenstein S, Zambon M, Yau E, Gorse GJ, Edelman R, Hayden FG, McElhaney JE, Neuzil KM, Nichol KL, Simoes EA, Wright PF, Sales VM. Comparison of the safety and immunogenicity of 2 respiratory syncytial virus (rsv) vaccines--nonadjuvanted vaccine or vaccine adjuvanted with alum--given concomitantly with influenza vaccine to high-risk elderly individuals. J Infect Dis. 2008 Nov 1;198(9):1317-26. doi: 10.1086/592168. PMID 18855558
- [Background] Widmer K, Griffin MR, Zhu Y, Williams JV, Talbot HK. Respiratory syncytial virus- and human metapneumovirus-associated emergency department and hospital burden in adults. Influenza Other Respir Viruses. 2014 May;8(3):347-52. doi: 10.1111/irv.12234. Epub 2014 Feb 7. PMID 24512531
- [Background] Lee N, Lui GC, Wong KT, Li TC, Tse EC, Chan JY, Yu J, Wong SS, Choi KW, Wong RY, Ngai KL, Hui DS, Chan PK. High morbidity and mortality in adults hospitalized for respiratory syncytial virus infections. Clin Infect Dis. 2013 Oct;57(8):1069-77. doi: 10.1093/cid/cit471. Epub 2013 Jul 21. PMID 23876395
- [Background] Zambon MC, Stockton JD, Clewley JP, Fleming DM. Contribution of influenza and respiratory syncytial virus to community cases of influenza-like illness: an observational study. Lancet. 2001 Oct 27;358(9291):1410-6. doi: 10.1016/s0140-6736(01)06528-x. PMID 11705487
- [Background] Sundaram ME, Meece JK, Sifakis F, Gasser RA Jr, Belongia EA. Medically attended respiratory syncytial virus infections in adults aged >/= 50 years: clinical characteristics and outcomes. Clin Infect Dis. 2014 Feb;58(3):342-9. doi: 10.1093/cid/cit767. Epub 2013 Nov 21. PMID 24265361
- [Background] Griffin MR, Coffey CS, Neuzil KM, Mitchel EF Jr, Wright PF, Edwards KM. Winter viruses: influenza- and respiratory syncytial virus-related morbidity in chronic lung disease. Arch Intern Med. 2002 Jun 10;162(11):1229-36. doi: 10.1001/archinte.162.11.1229. PMID 12038940
- [Background] Bianchini S, Silvestri E, Argentiero A, Fainardi V, Pisi G, Esposito S. Role of Respiratory Syncytial Virus in Pediatric Pneumonia. Microorganisms. 2020 Dec 21;8(12):2048. doi: 10.3390/microorganisms8122048. PMID 33371276
- [Background] Pneumonia Etiology Research for Child Health (PERCH) Study Group. Causes of severe pneumonia requiring hospital admission in children without HIV infection from Africa and Asia: the PERCH multi-country case-control study. Lancet. 2019 Aug 31;394(10200):757-779. doi: 10.1016/S0140-6736(19)30721-4. Epub 2019 Jun 27. PMID 31257127
- [Background] Loubet P, Voiriot G, Houhou-Fidouh N, Neuville M, Bouadma L, Lescure FX, Descamps D, Timsit JF, Yazdanpanah Y, Visseaux B. Impact of respiratory viruses in hospital-acquired pneumonia in the intensive care unit: A single-center retrospective study. J Clin Virol. 2017 Jun;91:52-57. doi: 10.1016/j.jcv.2017.04.001. Epub 2017 Apr 22. PMID 28494435
- [Background] Feddema JJ, Claassen E. Prevalence of viral respiratory infections amongst asthmatics: Results of a meta-regression analysis. Respir Med. 2020 Nov;173:106020. doi: 10.1016/j.rmed.2020.106020. Epub 2020 May 15. PMID 33190740
- [Background] Cilloniz C, Pericas JM, Rojas JR, Torres A. Severe Infections Due to Respiratory Viruses. Semin Respir Crit Care Med. 2022 Feb;43(1):60-74. doi: 10.1055/s-0041-1740982. Epub 2022 Feb 16. PMID 35172359
- [Background] Luyt CE. Virus diseases in ICU patients: a long time underestimated; but be aware of overestimation. Intensive Care Med. 2006 Jul;32(7):968-70. doi: 10.1007/s00134-006-0203-9. Epub 2006 May 24. No abstract available. PMID 16791659
- [Background] Sigurs N, Gustafsson PM, Bjarnason R, Lundberg F, Schmidt S, Sigurbergsson F, Kjellman B. Severe respiratory syncytial virus bronchiolitis in infancy and asthma and allergy at age 13. Am J Respir Crit Care Med. 2005 Jan 15;171(2):137-41. doi: 10.1164/rccm.200406-730OC. Epub 2004 Oct 29. PMID 15516534
- [Background] Stein RT, Sherrill D, Morgan WJ, Holberg CJ, Halonen M, Taussig LM, Wright AL, Martinez FD. Respiratory syncytial virus in early life and risk of wheeze and allergy by age 13 years. Lancet. 1999 Aug 14;354(9178):541-5. doi: 10.1016/S0140-6736(98)10321-5. PMID 10470697
- [Background] Beasley R, Coleman ED, Hermon Y, Holst PE, O'Donnell TV, Tobias M. Viral respiratory tract infection and exacerbations of asthma in adult patients. Thorax. 1988 Sep;43(9):679-83. doi: 10.1136/thx.43.9.679. PMID 3194873
- [Background] Gehlhar K, Bilitewski C, Reinitz-Rademacher K, Rohde G, Bufe A. Impaired virus-induced interferon-alpha2 release in adult asthmatic patients. Clin Exp Allergy. 2006 Mar;36(3):331-7. doi: 10.1111/j.1365-2222.2006.02450.x. PMID 16499644
- [Background] Grissell TV, Powell H, Shafren DR, Boyle MJ, Hensley MJ, Jones PD, Whitehead BF, Gibson PG. Interleukin-10 gene expression in acute virus-induced asthma. Am J Respir Crit Care Med. 2005 Aug 15;172(4):433-9. doi: 10.1164/rccm.200412-1621OC. Epub 2005 May 13. PMID 15894599
- [Background] van Scott MR, Justice JP, Bradfield JF, Enright E, Sigounas A, Sur S. IL-10 reduces Th2 cytokine production and eosinophilia but augments airway reactivity in allergic mice. Am J Physiol Lung Cell Mol Physiol. 2000 Apr;278(4):L667-74. doi: 10.1152/ajplung.2000.278.4.L667. PMID 10749743
- [Background] Hancock GE, Scheuer CA, Sierzega R, Pryharski KS, McBride JT, Watelet LF, Tebbey PW, Smith JD. Adaptive immune responses of patients with asthma to the attachment (G) glycoprotein of respiratory synctial virus. J Infect Dis. 2001 Dec 15;184(12):1589-93. doi: 10.1086/324583. PMID 11776949
- [Background] O'Sullivan S, Cormican L, Faul JL, Ichinohe S, Johnston SL, Burke CM, Poulter LW. Activated, cytotoxic CD8(+) T lymphocytes contribute to the pathology of asthma death. Am J Respir Crit Care Med. 2001 Aug 15;164(4):560-4. doi: 10.1164/ajrccm.164.4.2102018. PMID 11520715
- [Background] Coyle AJ, Erard F, Bertrand C, Walti S, Pircher H, Le Gros G. Virus-specific CD8+ cells can switch to interleukin 5 production and induce airway eosinophilia. J Exp Med. 1995 Mar 1;181(3):1229-33. doi: 10.1084/jem.181.3.1229. PMID 7869040
- [Background] Bjornsson E, Hjelm E, Janson C, Fridell E, Boman G. Serology of respiratory viruses in relation to asthma and bronchial hyperresponsiveness. Ups J Med Sci. 1996;101(2):159-68. doi: 10.3109/03009739609178920. PMID 8897706
- [Background] Douville RN, Bastien N, Li Y, Simons FE, HayGlass KT. Adult asthmatics display exaggerated IFNgamma responses to human metapneumovirus and respiratory syncytial virus. Biochem Cell Biol. 2007 Apr;85(2):252-8. doi: 10.1139/O07-005. PMID 17534407
- [Background] Hirose H, Matsuse H, Tsuchida T, Fukahori S, Fukushima C, Mizuta Y, Kohno S. Cytokine production from peripheral blood mononuclear cells of mite allergen-sensitized atopic adults stimulated with respiratory syncytial virus and mite allergen. Int Arch Allergy Immunol. 2008;146(2):149-55. doi: 10.1159/000113518. Epub 2008 Jan 18. PMID 18204281
- [Background] Lukacs NW, Tekkanat KK, Berlin A, Hogaboam CM, Miller A, Evanoff H, Lincoln P, Maassab H. Respiratory syncytial virus predisposes mice to augmented allergic airway responses via IL-13-mediated mechanisms. J Immunol. 2001 Jul 15;167(2):1060-5. doi: 10.4049/jimmunol.167.2.1060. PMID 11441116
- [Background] Johnson TR, Parker RA, Johnson JE, Graham BS. IL-13 is sufficient for respiratory syncytial virus G glycoprotein-induced eosinophilia after respiratory syncytial virus challenge. J Immunol. 2003 Feb 15;170(4):2037-45. doi: 10.4049/jimmunol.170.4.2037. PMID 12574374
- [Background] McLaughlin JM, Khan F, Begier E, Swerdlow DL, Jodar L, Falsey AR. Rates of Medically Attended RSV Among US Adults: A Systematic Review and Meta-analysis. Open Forum Infect Dis. 2022 Jun 17;9(7):ofac300. doi: 10.1093/ofid/ofac300. eCollection 2022 Jul. PMID 35873302
- [Background] Zhang Y, Sakthivel SK, Bramley A, Jain S, Haynes A, Chappell JD, Hymas W, Lenny N, Patel A, Qi C, Ampofo K, Arnold SR, Self WH, Williams DJ, Hillyard D, Anderson EJ, Grijalva CG, Zhu Y, Wunderink RG, Edwards KM, Pavia AT, McCullers JA, Erdman DD. Serology Enhances Molecular Diagnosis of Respiratory Virus Infections Other than Influenza in Children and Adults Hospitalized with Community-Acquired Pneumonia. J Clin Microbiol. 2016 Dec 28;55(1):79-89. doi: 10.1128/JCM.01701-16. Print 2017 Jan. PMID 27795341
- [Background] Vega JM, Badia X, Badiola C, Lopez-Vina A, Olaguibel JM, Picado C, Sastre J, Dal-Re R; Covalair Investigator Group. Validation of the Spanish version of the Asthma Control Test (ACT). J Asthma. 2007 Dec;44(10):867-72. doi: 10.1080/02770900701752615. PMID 18097865
- [Background] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Background] Dafauce L, Romero D, Carpio C, Barga P, Quirce S, Villasante C, Bravo MF, Alvarez-Sala R. Psycho-demographic profile in severe asthma and effect of emotional mood disorders and hyperventilation syndrome on quality of life. BMC Psychol. 2021 Jan 6;9(1):3. doi: 10.1186/s40359-020-00498-y. PMID 33407846
- [Background] Galan I, Rodriguez-Artalejo F, Tobias A, Diez-Ganan L, Gandarillas A, Zorrilla B. Clustering of behavior-related risk factors and its association with subjective health. Gac Sanit. 2005 Sep-Oct;19(5):370-8. doi: 10.1157/13080135. PMID 16242095
- [Background] Zeevat F, Luttjeboer J, Paulissen JHJ, van der Schans J, Beutels P, Boersma C, Postma MJ; RESCEU Investigators. Exploratory Analysis of the Economically Justifiable Price of a Hypothetical RSV Vaccine for Older Adults in the Netherlands and the United Kingdom. J Infect Dis. 2022 Aug 12;226(Suppl 1):S102-S109. doi: 10.1093/infdis/jiab118. PMID 34522947
- [Background] Falsey AR, Walsh EE, Esser MT, Shoemaker K, Yu L, Griffin MP. Respiratory syncytial virus-associated illness in adults with advanced chronic obstructive pulmonary disease and/or congestive heart failure. J Med Virol. 2019 Jan;91(1):65-71. doi: 10.1002/jmv.25285. Epub 2018 Sep 24. PMID 30132922
- See also: Access in June 2021 — http://www.cdc.gov/vaccines/vpd/pertussis/
- See also: Access in June 2021 — http://www.salute.gov.it/imgs/C_17_pubblicazioni_2571_allegato.pdf
- See also: Access in June 2021 — http://www.fhi.no/sv/vaksine/voksenvaksinasjon/oversikt-anbefalte-vaksiner-for-voksne/
- See also: Access in June 2021 — https://goldcopd.org/wp-content/uploads/2020/11/GOLD-REPORT-2021-v1.1-25Nov20_WMV.pdf
- See also: June 2022 — https://ginasthma.org/wp-content/uploads/2022/07/GINA-Main-Report-2022-FINAL-22-07-01-WMS.pdf
- See also: 2022 — https://pnsd.sanidad.gob.es/profesionales/publicaciones/catalogo/catalogoPNSD/publicaciones/pdf/2022_Technical_Report_Alcohol_2021.pdf